CLINICAL TRIAL: NCT03657459
Title: Danger Signs of Worsening Heart Failure and Self-Management of Danger Signs: The Effects of Video Education
Brief Title: Danger Signs in Heart Failure- Effects of Video Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Wellflix, Inc. (Unknown)
Responsible Party: Principal Investigator, Nancy M. Albert, Ph.D., Assocaite Chief Nursing Officer-Resaerch and Senior Nurse Scientist, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-442
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Results first posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; With Decompensation
Keywords: video education; self care management; symptom recognition
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomized, controlled prospective trial
Who Masked: Care Provider, Investigator
Masking Description: Documentation of enrollment will not include group assignment Investigator will be blinded from group assignment via a separate excel file with that detail
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual care group (No Intervention): Usual care consists of patient's receiving a Heart Failure Handbook before hospital discharge + verbal education delivered by multiple care providers (including a group education class at 1 site). The handbook is consistent; however, verbal education may vary between care providers based on their knowledge and time available, and perceived patient needs
- video education group (Active Comparator): Will receive usual care, plus will watch 2 short Wellflix, Inc. Danger Signs of Heart Failure videos (via iPAD) on dyspnea, fatigue + a Danger Sign "edema" video, when applicable. Each video describes how to recognize if the sign/symptom is new or worsening and how to self-manage at home (via diet, fluid management and activity instructions)
  Interventions: Behavioral: Danger Signs of Heart Failure Videos

INTERVENTIONS:
Behavioral: Danger Signs of Heart Failure Videos — Short (under 3 minutes each) videos on (a) recognition of dyspnea, fatigue and edema and (b) self-management of each (based on diet, fluid management and activities) that reflect patient behaviors
  Arms: video education group

SUMMARY:
Lack of recognition of HF danger signs and lack of understanding of how to control and minimize danger signs could lead to their escalation and prompt all-cause and HF-related health care resource utilization (HCRU). Investigators hypothesize that patients must understand HF danger signs to have self-confidence in recognizing them and in taking steps to minimize or eliminate their occurrence post hospital discharge. Investigators will determine if video education in HF danger signs recognition and control prior to discharge (and post-discharge) reduces all-cause and HF-related HCRU.

DETAILED DESCRIPTION:
The most frequently cited danger signs of heart failure (HF) are new onset or worsening of fatigue, dyspnea and edema. In previous research, patients did not recognize worsening HF, due to 3 primary reasons: (1) danger signs were non-specific and misinterpreted as stress, an external force or another comorbidity, (2) danger signs were unrecognized due to the subtle nature of worsening status, or (3) when patients eliminated or minimized activities that prompted danger signs, they interpreted the results as improvement in status. Lack of recognition of HF danger signs and lack of understanding of how to control and minimize danger signs could lead to their escalation and prompt all-cause and HF-related health care resource utilization (HCRU). Investigators hypothesize that patients must understand HF danger signs to have self-confidence in recognizing them and in taking steps to minimize or eliminate their occurrence post hospital discharge. The purposes of this trial are to determine if video education in HF danger signs recognition and control prior to discharge (and post-discharge) reduces all-cause and HF-related health care resource utilization. The intervention will be administered during hospitalization, and patients and family members will receive a link to a website and a DVD to review videos as often as desired post-discharge. The primary end-point is 30-day HF-related hospitalization. 732 patients (658 + 10% attrition) with decompensated HF will be enrolled from multiple hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Not referred for cardiac transplantation or ventricular assist device placement during the index hospitalization,
* Cognitively intact and able to view videos (adequate eyesight and hearing) with correction, if needed,
* Discharge to home, assisted living facility or to a family member's home and can control dietary sodium and fluids as needed,
* Willing to participate; which may require up to three (3) follow-up telephone calls post-discharge.

Exclusion Criteria:

* Chart documented psychiatric or cognitive conditions that limit ability to understand video content or adhere to self-care recommendations (Alzheimer's condition, dementia, schizophrenia, other neurological history that impairs memory or concentration),
* Plans to discharge to skilled nursing facility or hospice care,
* Receiving home hospice or palliative care; or has a medical condition reflecting less than 1 year of survival (cachexia, end stage liver disease or cancer or non-ambulatory New York Heart Association functional class IV HF),
* Hospitalized but at admission, in New York Heart Association functional class I or II HF
* Post-cardiac transplantation or ventricular assist device placement,
* Currently enrolled in another experimental HF research study,
* Chronic renal failure and receiving chronic hemodialysis therapy for an estimated glomerular filtration rate < 15 mL/minute/1.73 m2,
* A non-traditional form of HF (hypertrophic or restrictive forms of cardiomyopathy, congenital heart disease or Takotsubo cardiomyopathy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Please answer each question as it applies to you.
  Sex: 0.______ Male 1.______ Female
Enrollment: 746 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NANCY M. ALBERT, PhD, Principal Investigator — The Cleveland Clinic
Locations (8):
- United States (8):
  - Medical Center Navicent Health, Macon, Georgia
  - Cleveland Clinic Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic main campus, Cleveland, Ohio
  - Cleveland Clinic Marymount Hospital, Garfield Heights, Ohio
  - Cleveland Clinic Hillcrest Hospital, Mayfield Heights, Ohio
  - Cleveland Clinic Medina Hospital, Medina, Ohio
  - Cleveland Clinic South Pointe Hospital, Warrensville Heights, Ohio
  - WellSpan Health, York, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No plans to share individual data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients with decompensated HF, with preserved or reduced ejection fraction when hospitalized and New York Heart Association FC III or ambulatory IV symptoms, were recruited for this study between July 2018 to November 2020.
Pre-assignment Details: In total, 746 patients started/completed study (377 patients randomized to usual care and 369 intervention).
Groups:
- Video Education Group: Will receive usual care, plus will watch 2 short Wellflix, Inc. Danger Signs of Heart Failure videos (via iPAD) on dyspnea, fatigue + a Danger Sign "edema" video, when applicable. Each video describes how to recognize if the sign/symptom is new or worsening and how to self-manage at home (via diet, fluid management and activity instructions)
  Danger Signs of Heart Failure Videos: Short (under 3 minutes each) videos on (a) recognition of dyspnea, fatigue and edema and (b) self-management of each (based on diet, fluid management and activities)
Period: Overall Study
Arm/Group | Usual Care Group | Video Education Group
Started | 377 | 369
Completed | 377 | 369
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Group | Video Education Group | Total
Number analyzed (Participants) | 377 | 369 | 746
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (12.5) | 67.7 (12.3) | 68.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 179 | 329
  Male | 227 | 190 | 417
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 116 | 118 | 234
  White | 253 | 243 | 496
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 377 | 369 | 746
Marital status [Count of Participants; unit: Participants]
  Single | 69 | 66 | 135
  Married, living with partner | 177 | 170 | 347
  Divorced/separated/widowed | 112 | 98 | 210
  Living with child or another person not a spouse or partner | 19 | 35 | 54
Someone who supports you [Count of Participants; unit: Participants]
  No, not needed | 18 | 16 | 34
  No, no supporter available | 18 | 14 | 32
  Yes, have a support person | 340 | 339 | 679
  Missing survey response | 1 | 0 | 1
Someone to confide in [Count of Participants; unit: Participants]
  No | 15 | 11 | 26
  Yes | 362 | 358 | 720
Highest level of education completed [Count of Participants; unit: Participants]
  High school or less | 205 | 204 | 409
  Some college | 86 | 72 | 158
  Bachelor/Associate/Professional degree | 57 | 62 | 119
  Master/Doctoral degree | 28 | 30 | 58
  Missing survey response | 1 | 1 | 2
Employment status [Count of Participants; unit: Participants]
  Employed full or part-time outside home | 40 | 53 | 93
  Unemployed by choice or homemaker | 17 | 14 | 31
  Sick leave or disability or retired due to HF | 84 | 91 | 175
  Retired, not due to HF | 225 | 202 | 427
  Other | 11 | 9 | 20
Consider how well you live on income [Count of Participants; unit: Participants]
  Comfortable, have more than enough to make ends meet | 99 | 125 | 224
  Have enough to make ends meet | 179 | 137 | 316
  Do not have enough to make ends meet | 96 | 107 | 203
  Missing survey response | 3 | 0 | 3
BMI [Median (Inter-Quartile Range); unit: Kg/m2] — measures the ratio of height to weight to estimate the amount of body fat a person has. BMI is calculated by using weight in kilograms (kg) divided by the square of height in meters (m2) [kg/m2].
  Kg/m2 | 32.2 [26.0 to 38.9] | 31.5 [25.8 to 38.6] | 31.9 [25.9 to 38.8]
Insurance [Count of Participants; unit: Participants]
  Government | 197 | 196 | 393
  Commercial | 39 | 30 | 69
  HMO | 38 | 38 | 76
  None | 8 | 9 | 17
  Government and commercial | 40 | 42 | 82
  Government and HMO | 55 | 54 | 109
How far away in miles is your home to the office/clinic? [Count of Participants; unit: Participants]
  Under 5 miles | 96 | 66 | 162
  Over 5 miles but under 15 miles | 114 | 127 | 241
  15 miles or over 20 minutes | 144 | 157 | 301
  I have not seen a HF medical provider in >1 year | 22 | 17 | 39
  Do not know the distance | 1 | 1 | 2
  Missing survey response | 0 | 1 | 1
How far away in miles is your home to the hospital [Count of Participants; unit: Participants]
  Under 5 miles | 125 | 112 | 237
  Over 5 miles but under 15 miles | 147 | 140 | 287
  15 miles or over 20 minutes | 100 | 114 | 214
  I have not seen a HF medical provider in >1 year | 3 | 2 | 5
  Do not know the distance | 2 | 1 | 3
In general would you say your health is [Count of Participants; unit: Participants]
  Excellent | 1 | 1 | 2
  Very good | 18 | 16 | 34
  Good | 109 | 93 | 202
  Fair | 158 | 154 | 312
  Poor | 90 | 105 | 195
  Missing survey response | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HF-related Healthcare Resource Utilization (HCRU)
Description: Number of participants post-discharge with HF-related healthcare resource utilization including hospitalization, emergency department (ED) visits, death, or cardiac transplant within 30 days of discharge.
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 64 | 59

2. Secondary Outcome: Number of Participants With HF-related Hospitalization
Description: Total number of participants post-discharge with HF-related hospitalization
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 52 | 51

3. Secondary Outcome: Number of Participants With HF-related ED Visits
Description: Number of participants with post-discharge HF-related ED visits
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 40 | 36

4. Secondary Outcome: Number of Participants With HF-related Death
Description: Number of participants post-discharge with HF-related death
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 5 | 4

5. Secondary Outcome: Number of Participants With HF-related Healthcare Resource Utilization (HCRU)
Description: Number of participants post-discharge with HF-related healthcare resource utilization including hospitalization, emergency department (ED) visits, death, or cardiac transplant within 90 days of discharge.
Time Frame: up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 93 | 102

6. Secondary Outcome: Number of Participants With HF-related Hospitalization
Description: Number of participants post-discharge with HF-related hospitalization
Time Frame: up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 87 | 95

7. Secondary Outcome: Number of Participants With HF-related ED Visit
Description: Number of participants post-discharge with HF-related ED visit
Time Frame: up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 63 | 70

8. Secondary Outcome: Number of Participants With HF-related Death
Description: Number of participants post-discharge with HF-related death
Time Frame: up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 12 | 11

9. Secondary Outcome: Number of Participants With HF-related Healthcare Resource Utilization (HCRU)
Description: Number of participants post-discharge with HF-related healthcare resource utilization including hospitalization, emergency department (ED) visits, death, or cardiac transplant within 180 days of discharge.
Time Frame: up to 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 111 | 135

10. Secondary Outcome: Number of Participants With HF-related Hospitalization
Description: Number of participants post-discharge with HF-related hospitalization
Time Frame: up to 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 104 | 128

11. Secondary Outcome: Number of Participants With HF-related ED Visit
Description: Number of participants post-discharge with HF-related ED visit
Time Frame: up to 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 73 | 91

12. Secondary Outcome: Number of Participants With HF-related Death
Description: Number of participants post-discharge with HF-related death
Time Frame: up to 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 15 | 14

13. Secondary Outcome: Number of Participants With All-cause Healthcare Resource Utilization (HCRU)
Description: Number of participants post-discharge with all-cause healthcare resource utilization including hospitalization, emergency department (ED) visits, death, or cardiac transplant within 30 days of discharge.
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 124 | 130

14. Secondary Outcome: Number of Participants With All-cause Hospitalization
Description: Number of participants post-discharge with all-cause hospitalization
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 75 | 78

15. Secondary Outcome: Number of Participants With All-cause ED Visits
Description: Number of participants with post-discharge all-cause ED visits
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 79 | 84

16. Secondary Outcome: Number of Participants With All-cause Death
Description: Number of participants post-discharge with all-cause deaths
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 13 | 11

17. Secondary Outcome: Number of Participants With All-cause Healthcare Resource Utilization (HCRU)
Description: Number of participants post-discharge with all-cause healthcare resource utilization including hospitalization, emergency department (ED) visits, death, or cardiac transplant within 90 days of discharge.
Time Frame: up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 194 | 194

18. Secondary Outcome: Number of Participants With All-cause Hospitalization
Description: Number of participants with post-discharge all-cause hospitalization
Time Frame: up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 148 | 134

19. Secondary Outcome: Number of Participants With All-cause ED Visits
Description: Number of participants post-discharge with all-cause ED visits
Time Frame: up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 132 | 134

20. Secondary Outcome: Number of Participants With All-cause Death
Description: Number of participants post-discharge with all-cause death
Time Frame: up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 30 | 22

21. Secondary Outcome: Number of Participants With All-cause Healthcare Resource Utilization (HCRU)
Description: Number of participants post-discharge with all-cause healthcare resource utilization including hospitalization, emergency department (ED) visits, death, or cardiac transplant within 180 days of discharge.
Time Frame: up to 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 232 | 242

22. Secondary Outcome: Number of Participants With All-cause Hospitalization
Description: Number of participants post-discharge with all-cause hospitalization
Time Frame: up to 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 195 | 188

23. Secondary Outcome: All-cause ED Visits at 180 Days
Description: Number of participants post-discharge with all-cause ED visits
Time Frame: up to 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 160 | 179
Statistical Analysis 1: Comparison: Usual Care Group vs Video Education Group; Test type: Superiority; p = 0.0096, Chi-squared; Pearsons Chi Square

24. Secondary Outcome: All-cause Death at 180 Days Post Discharge
Description: Number of participants post-discharge with all-cause death
Time Frame: up to 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 377 | 369
Participants | 42 | 40
Statistical Analysis 1: Comparison: Usual Care Group vs Video Education Group; Test type: Superiority; p = 0.90, Chi-squared — no adjustment; Pearson Chi-square

25. Secondary Outcome: Functional Status Using the Duke Acrivity Status Index Scale at 30 Days Post Discharge
Description: Duke Activity Status Index (DASI) score at 30 days. Patients completed the DASI, a 12-item questionnaire using a Likert-like scale that determines a patient's ability to participate in daily self-care activities including ambulation, housework, yard work, sexual relations, and recreational activities. A total score reflects functional status based on responses. The full range of scores is 0 (most severe functional impairment) to 58.2 (no functional impairment). There is no established cut-point for this scale. Positive, higher scores reflect a positive and better functional status.
Time Frame: up to 30 days
Population: The number analyzed in both groups was lower than the number enrolled. This is due to the research team being unable to contact some patients by phone for study follow-up or the patient was deceased (medical record chart review).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Video Education Group: Will receive usual care, plus will watch Wellflix, Inc. Danger Signs of Heart Failure videos (via iPAD) on dyspnea, fatigue + a Danger Sign "edema" video, when applicable. Each video describes how to recognize if the sign/symptom is new or worsening and how to self-manage at home (via diet, fluid management and activity instructions)
  Danger Signs of Heart Failure Videos: Short (under 3 minutes each) videos on (a) recognition of dyspnea, fatigue and edema and (b) self-management of each (based on diet, fluid management and activities)
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 334 | 330
score on a scale | 17.2 (11.2) | 18.2 (11.6)

26. Secondary Outcome: Dyspnea at 30 Days Post Discharge
Description: PROMIS® Dyspnea Functional Limitations - Short Form 10a was used. It is a 10-item tool that measures dyspnea by asking 10 questions about the difficulty in completing activities in the past 7 days. Responses range from "0 = no difficulty" to "3 = much difficulty" and there is an option for "I did not do this in the past 7 days" - there were 5 response options in total. Minimum and maximum raw scores are 0-30. PROMIS T scores are standardized with scores around 50 (standard deviation of 10) equating to normal/average levels and scores above or below equating to heightening or lessening of the variable being measured. A 5 point change in score is considered significant. A table is used to translate the total raw score to T score for each participant.
Time Frame: 30 days
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 321 | 319
score on a scale | 46.1 (8.5) | 45.8 (8.5)

27. Secondary Outcome: Fatigue at 30 Days Post Discharge
Description: 10-item Fatigue Assessment Scale from baseline. The Fatigue Assessment Scale is a valid, reliable 10-item scale evaluating symptoms of chronic fatigue. It uses Likert-type response options ranging from 1 ("never") to 5 ("always"), with some items reverse scored. Total scores range from 10 (lowest level of fatigue) to 50 (highest level of fatigue).
Time Frame: to 30 days
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 322 | 320
score on a scale | 23.8 (8.5) | 23.3 (8.4)

28. Secondary Outcome: Self-efficacy for Managing Symptoms at 30 Days Post Discharge
Description: PROMIS Self-Efficacy for Managing Symptoms Short form 8a for managing symptoms, from baseline. 8-item tool that ranges from 'I am not at all confident' to 'I am very confident" - higher scores equals higher self-efficacy. A mean score of 50 is the average score in the general population of U.S. with standard deviation of 10. A table is used to translate the total raw score to T score for each participant. The T score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. Higher scores (above 50) reflect better than average self-efficacy
Time Frame: 30 days
Population: The number analyzed in both groups was lower than the number enrolled. This is due to the research team being unable to contact some patients by phone for study follow-up or the patient was deceased (medical record).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care Group | Video Education Group
Number analyzed (Participants) | 322 | 319
score on a scale | 42.9 (8.4) | 43.4 (7.8)

29. Secondary Outcome: Intervention Group Only- All-cause Events Based on Dichotomous Metric of Viewing the Video at Home (Never vs 1+)
Description: Among intervention group participants, total number of all-cause events within 30 days of discharge, based on the number of times the patient watched the video education. Participant responses are grouped into two categories: Never watched vs. 1 or more times
Time Frame: 30 days
Population: The number analyzed (n=304) was lower than the number enrolled due to inability to contact some patients by phone for study follow-up or the patient was deceased (as a note, this info was not available in the medical record).
Measure: Count of Participants; unit: Participants
Groups:
- Video Education Group - Never Watched Video at Home: Video delivered and watched during hospitalization but never watched at home
- Video Education Group - Watched 1+ Time at Home: Video delivered and watched during hospitalization, and watched 1+ or more times at home
Arm/Group | Video Education Group - Never Watched Video at Home | Video Education Group - Watched 1+ Time at Home
Number analyzed (Participants) | 227 | 77
Participants | 76 | 25

30. Secondary Outcome: Intervention Group Only; Number of All-cause Events Based on Dichotomous Outcome of Family Member Viewing Educational Video After Hospital Discharge (Yes vs no)
Description: Total number of participants (video education group only), comparison of all-cause events within 30 days of discharge, based on family members watching the educational videos after the hospital (Yes/No).
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Video Education Group - NO, Family Never Watched: Video education group but family member never reviewed video content
- Video Education Group - YES, Family Watched: Video education group and family member reviewed video content at least 1 time
Arm/Group | Video Education Group - NO, Family Never Watched | Video Education Group - YES, Family Watched
Number analyzed (Participants) | 272 | 32
Participants | 94 | 7

ADVERSE EVENTS:
Time Frame: Adverse events recorded for this study were NON-treatment-related. Patient charts were monitored at 180 days (6 months) and considered to be non-direct patient outcomes becasue of the nature of participants medical condition, in general.
Description: Adverse events were NON-treatment-related as the intervention was video education. The IRB approved this study as minimal risk and adverse events were NOT collected or recorded except those believed to be important indirect (no direct) heart failure and all-cause 180 day outcomes (death, emaergency department visits and hospitalizations). Patient charts were monitored for the above outcomes at180 days (6 months).
Groups:
- Video Education Group: Will receive usual care, plus will watch short videos from Wellflix, Inc.: 1) "Danger Signs of Heart Failure" videos (via iPAD) on dyspnea and fatigue; and 2) "Danger Signs edema" video. Each video describes how to recognize if the patient's signs/symptoms are new or worsening and how to self-manage at home via diet, fluid management, and physical activity instructions.
  Danger Signs of Heart Failure Videos are short videos (less than 3 minutes each). The videos contain educational information on (a) recognition of dyspnea, fatigue, and edema; and (b) self-management (based on diet, fluid management, and activities)
Arm/Group | Usual Care Group | Video Education Group
All-Cause Mortality (participants affected / at risk) | 42/377 | 40/369
Serious Adverse Events (participants affected / at risk) | 232/377 | 242/369
Other Adverse Events (participants affected / at risk) | 0/377 | 0/369
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care Group (N=377) | Video Education Group (N=369)
All-cause 180 day emergency department, hospitalization, transplant/left ventricular assist device o (Cardiac disorders) | 232 | 242 — Events were considered non-direct in relation to the education video as education is an INDIRECT effect of all-cuase related outcomes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT03657459/Prot_SAP_000.pdf